CLINICAL TRIAL: NCT04799067
Title: Hyperkalaemia Prevalence, Recurrence and Treatment in Haemodialysis: A Prospective Multi-centre Cohort Study
Brief Title: Hyperkalaemia Prevalence, Recurrence and Treatment in Haemodialysis
Acronym: PRECEDE-K
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9480R00033; No secondary ID yet (Other: No secondary ID yet)
Record Dates: First submitted 2021-02-24; First posted 2021-03-16 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Hyperkalemia; Hemodialysis; Water-Electrolyte Imbalance
Keywords: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia; Water-Electrolyte Imbalance | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational study — no study drug involved, observational study.

SUMMARY:
The objective of this study is to evaluate the prevalence and recurrence of Hyperkalaemia (HK) in Chinese HD patients and to understand the treatment pattern of HK in China.

DETAILED DESCRIPTION:
This is a prospective, cohort study. This study will include approximate 600 End Stage Renal Disease (ESRD) patients receiving Haemodialysis (HD) treatment twice a week or thrice a week.

The assessments at enrolment and in follow-up are summarized as follow:

Enrolment - Patients will be in Long Interdialytic interval (LIDI) at enrolment (V1). Demographic characteristics, medical history, etiology of ESRD, concomitant medications, dialysis vintage, an electrocardiogram (ECG), a pre-dialysis serum potassium measurement and a post- dialysis serum potassium measurement, blood routine, blood gas analysis and other blood biochemistry measurements, etc., will be obtained.

Follow-up - Potassium measurements, including pre-dialysis potassium measurements at LIDI once every month (V3-V8), pre-dialysis potassium at SIDI during the first week (V2) for patients in HD thrice a week specifically, will be obtained. Concomitant medications, blood routine, blood gas analysis and other blood biochemistry measurements, etc., will be obtained

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged ≥ 18 years at the time of signing the informed consent.
2. Patients with ESRD and on haemodialysis (HD)
3. The HD treatment frequency is ≥2 sessions per week
4. Capable of giving signed informed consent

Exclusion Criteria:

1. Acute kidney injury
2. Expected to receive renal transplantation within 6 months
3. Intracranial haemorrhage or elevated intracranial pressure within one month before enrolment
4. Shock that cannot be corrected by drugs within one month before enrolment
5. Failure to establish vascular access
6. Has been receiving peritoneal dialysis
7. Not suitable for this study judged by investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ESRD patients receiving HD treatment twice a week or thrice a week.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Proportion of patients experiencing any HK at the study enrolment or during a 24-week follow-up | up to 24 weeks
  Proportion of patients experiencing any HK (defined as serum potassium > 5.0 mmol/L) at the study enrolment or during a 24-week follow-up

SECONDARY OUTCOMES:
Proportion of patients experiencing HK recurrence within 1, 2, 3, 4, 5 or 6 months (if applicable) during a 24-week follow-up including enrolment assessment | up to 24 weeks
  Proportion of patients experiencing HK recurrence (defined as any HK event after the first HK event) within 1, 2, 3, 4, 5 or 6 months (if applicable) during a 24-week follow-up including enrolment assessment. A HK event is defined as any serum K+> 5.0 mmol/L within an interdialytic interval, which is usually two to three days.
Proportion of patients with 2, 3, 4, 5, 6 or more than 6 events of HK during a 24-week follow-up including enrolment assessment | up to 24 weeks
  Proportion of patients with 2, 3, 4, 5, 6 or more than 6 events of HK during a 24-week follow-up including enrolment assessment
Intradialytic potassium shift at LIDI during the first week after patient enrolment | up to 1 week
  Intradialytic potassium shift (defined as the difference between pre- and post-dialysis K+)at LIDI during the first week after patient enrolment
Serum K+ at LIDI and SIDI in patients receiving HD thrice a week during the first week after patient enrolment | up to 1 week
  Serum K+ at LIDI and SIDI in patients receiving HD thrice a week during the first week after patient enrolment
Proportion of HK patients treated with any potassium binders and specific proportion of each potassium binder respectively during the 24-week follow up period | up to 24 weeks
  Proportion of HK patients treated with any potassium binders including sodium polystyrene sulfonate ( calcium polystyrene sulfonate (CPS) or sodium zirconium cyclosilicate (SZC), and specific proportion of each potassium binder respectively during the 24-week follow up period
Proportion of HK events treated with any potassium binders including SPS, CPS or SZC among total number of HK events during the 24-week follow up period | up to 24 weeks
  Proportion of HK events treated with any potassium binders among total number of HK events during the 24-week follow up period
Mean daily dose of SPS, CPS or SZC in patients treated with any potassium binder | up to 24 weeks
  Mean daily dose of SPS, CPS or SZC in patients treated with any potassium binder
Duration of the treatment of SPS, CPS or SZC in patients treated with any potassium binders | up to 24 weeks
  Duration of the treatment of SPS, CPS or SZC in patients treated with any potassium binders

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Shenzhen, Guangdong
  - Research Site, Shijiazhuang, Hebei
  - Research Site, Taihe, Hubei
  - Research Site, Nanchang, Jiangxi
  - Research Site, Shenyang, Liaoning
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Taiyuan, Shanxi
  - Research Site, Yangquan, Shanxi
  - Research Site, Ningbo, Zhejiang
  - Research Site, Wenzhou, Zhejiang

REFERENCES:
- [Derived] Jin H, Lu R, Zhang L, Yao L, Shao G, Zuo L, Qin S, Zhang X, Zhang Q, Yu W, Luo Q, Ren Y, Peng H, Xiao J, Yang Q, Chen Q, Shi Y, Ni Z. Hyperkalemia burden and treatment patterns in Chinese patients on hemodialysis: final analysis of a prospective multicenter cohort study (PRECEDE-K). Ren Fail. 2024 Dec;46(2):2384585. doi: 10.1080/0886022X.2024.2384585. Epub 2024 Sep 9. PMID 39252179
- [Derived] Ni Z, Jin H, Lu R, Zhang L, Yao L, Shao G, Zuo L, Qin S, Zhang X, Zhang Q, Yu W, Luo Q, Ren Y, Peng H, Xiao J, Yang Q, Chen Q, Shi Y; PRECEDE-K study group. Hyperkalaemia prevalence and dialysis patterns in Chinese patients on haemodialysis: an interim analysis of a prospective cohort study (PRECEDE-K). BMC Nephrol. 2023 Aug 9;24(1):233. doi: 10.1186/s12882-023-03261-8. PMID 37559023
- [Derived] Ni Z, Jin H, Lu R, Zuo L, Yu W, Ren Y, Yang Q, Xiao J, Zhang Q, Zhang L, Zhang X, Chen Q, Chen C, Shao G, Luo Q, Yao L, Qin S, Peng H, Zhao Q; PRECEDE-K Study group. Hyperkalaemia prevalence, recurrence and treatment in patients on haemodialysis in China: protocol for a prospective multicentre cohort study (PRECEDE-K). BMJ Open. 2021 Dec 22;11(12):e055770. doi: 10.1136/bmjopen-2021-055770. PMID 34937724
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480R00033&attachmentIdentifier=68e349a6-0176-4b00-b137-4af8956d8d35&fileName=D9480R00033_redacted_CSR_Synopsis.pdf&versionIdentifier=